CLINICAL TRIAL: NCT00382577
Title: A Randomized, Double-blind, Two Period, Crossover Study to Evaluate the Effects of a Single Dose of Itopride 200 mg on Esophageal and Gastric pH and Reflux in Patients With Heartburn
Brief Title: Efficacy and Safety of Itopride vs Placebo in Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ITOLES06-01
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — itopride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Itopride
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of itopride in patients with heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy males and females aged 18-70, with at least 3 episodes of heartburn or acid regurgitation per week.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
24-hour pH Monitoring | after 5 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Philip, Jr. B. Miner, M.D., Principal Investigator — The Oklahoma Foundation for Digestive Research
Locations (1):
- The Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma, United States